CLINICAL TRIAL: NCT04513470
Title: A Multi-Center, Open-Label Study, Evaluating Safety of Allocetra-OTS for the Prevention of Organ-Failure Deterioration in Severe Patients With COVID-19 and Respiratory Dysfunction
Brief Title: Allocetra-OTS in COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Mevorach Dror, Professor & Head, Department of Internal Medicine B; Head, Rheumatology Research Center, Hadassah and the Hebrew University Medical School, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DM003
Record Dates: First submitted 2020-08-10; First posted 2020-08-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 (Experimental): Five subjects, male or female > 18 and < 80-year-old diagnosed with respiratory dysfunction and COVID-19, as defined in the Eligibility Criteria, and treated with a single intravenous dose of Allocetra-OTS investigational product as detailed in the Interventions section.
  Interventions: Biological: Allocetra-OTS

INTERVENTIONS:
Biological: Allocetra-OTS — Allocetra-OTS is a cell-based therapeutic composed of donor early apoptotic cells, comprising allogeneic mononuclear enriched cell suspension with at least 40% early apoptotic cells. The suspension is prepared with Ringer's lactate solution and administered IV. It is stored at 2-8°C until 20+25 minutes before infusion and at room temperature thereafter. Each dose contains 140x10E6 ± 20% cells/ kg of recipient body weight (at screening) in a total volume of 375 mL in a transfer pack that undergoes irradiation and is administered via an adjusted filter using a volumetric pump, at a starting rate of 48 mL/hour with a gradual increase every 15-25 minutes of 15 mL/hour to a maximal rate of 102 mL/hour. The study intervention should be completed within 72 hours of completing the manufacturing process. During product administration, no other IV fluids such as Ringer's lactate or normal saline will be given in parallel unless medically indicated due to volume depletion.

SUMMARY:
This is a multi-center, open-label study evaluating the safety of Allocetra-OTS, in 5 subjects with severe COVID-19 and respiratory dysfunction. Subjects, who will be identified as suffering from COVID-19, will be recruited.

After signing an informed consent by the patient and, within 24+6 hours following the time of eligibility (time 0), on Day 1, eligible recipient subjects will receive single intravenous (IV) administration of investigational product as described below.

Subjects will be hospitalized for COVID-19, and later as medically indicated. Following investigational product (IP) administration (Day 1), subjects will be followed for efficacy and safety assessments through 28 days.

DETAILED DESCRIPTION:
Study Rationale

COVID-19, the name given to the clinical syndrome associated with the newly recognized virus severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has become pandemic with a mortality estimated based on reports from China between 1-3% and complications among hospitalized patients leading to up to 15-25% admissions to the Intensive Care Unit (ICU). The clinical presentation includes both upper and lower respiratory tract infection, but patients may also be asymptomatic.

The term "cytokine storm" calls up vivid images of an immune system gone awry and an inflammatory response flaring out of control. The term has captured the attention of the public and the scientific community alike and is increasingly being used in both the popular media and the scientific literature. Indeed, a few publications have indicated an important part of the complications in COVID-19 are related to a cytokine storm.

In that regard, the investigators have recently completed a successful phase 1b clinical trial of immune-modulation in patients with sepsis (NCT03925857).

Taken together, in patients with moderate to severe COVID-19, there may be a comparable underlying immunological mechanism of action that may be similar to the one that was recently shown by us in sepsis, which is a hyper-inflammatory pathway associated with increased death. 40 previous trials using monoclonal antibodies against a single cytokine in septic patients have failed in sepsis pointing out that there is a need to modify the cytokine storm rather than treating with a single anti-cytokine.

This solution is provided by Allocetra-OTS, which targets macrophages and dendritic cells that produce most of the cytokine storm.

Study Design This is a multi-center, open-label study evaluating the safety of Allocetra-OTS, in five subjects with severe COVID-19 and respiratory dysfunction. Subjects, who will be identified as suffering from COVID-19, will be recruited.

After signing an informed consent by the patient and, within 24+6 hours following the time of eligibility (time 0), on Day 1, eligible recipient subjects will receive single intravenous (IV) administration of investigational product as described below:

● Allocetra-OTS treatment at 140 x 106 ±20% cells/kg body weight (screening body weight) in 375 mL of Ringer's lactate solution.

Subjects will be followed for efficacy and safety assessments over 28 days following investigational product administration.

Subjects will be hospitalized for COVID-19, and later as medically indicated. Following IP administration (Day 1), subjects will be followed for efficacy and safety assessments through 28 days. The number of visits for subjects participating in this study will be on Days 3, 5, 7, 14, and 28.

Study Intervention, Route of Administration, and Dosage Form Allocetra-OTS is a cell-based therapeutic composed of donor early apoptotic cells.

Patient Classification [National Institutes of Health (NIH)]- www.covid19treatmentguidelines.nih.gov/overview/management-of-covid-19/

In general, adults with COVID-19 can be grouped into the following severity of illness categories:

* Asymptomatic or Pre-symptomatic Infection: Individuals who test positive for SARS-CoV-2 by virologic testing using a molecular diagnostic (e.g., polymerase chain reaction) or antigen test, but have no symptoms.
* Mild Illness: Individuals who have any of the various signs and symptoms of COVID-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain) without shortness of breath, dyspnea, or abnormal chest imaging.
* Moderate Illness: Individuals who have evidence of lower respiratory disease by clinical assessment or imaging and saturation of oxygen (SpO2) ≥94% on room air at sea level.
* Severe Illness: Individuals who have respiratory frequency >30 breaths per minute, SpO2 <94% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mmHg, or lung infiltrates >50%
* Critical Illness: Individuals who have respiratory failure, septic shock, and/or multiple organ dysfunction.

Standard of Care (SOC) The SOC for COVID-19 will be according to institutional standards. Institutional SOC may include Clexane, anti-viral agents such as Remdesivir, Dexamethasone, or other agents.

Concomitant Medications Prohibited medications: Significant immune-suppressing agents including Azathioprine, Cyclosporine, Cyclophosphamide, and any biological treatment.

Concomitant Medical Conditions Apart from patients with a tumor or end-stage organ condition, chronic diseases like cardiovascular or diabetes are allowed.

ELIGIBILITY:
Inclusion Criteria:

Five subjects, male or female > 18 and < 80-year-old diagnosed with respiratory dysfunction and COVID-19, as defined below:

1. Laboratory confirmation of SARS-CoV-2 infection by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source.
2. Patients classified as severe according to NIH severity classification.
3. All patients will be treated by treating physicians with subcutaneous (S.C.) Clexane, at a minimal dose of 40 mg a day

Exclusion Criteria:

1. Pregnancy, lactation, and childbearing potential woman who are not willing to use acceptable contraceptives measures for the entire study duration.
2. Combined with other organ failures (need organ support not including respirator), including Stage 4 severe chronic kidney disease or requiring dialysis (i.e. estimated glomerular filtration rate (eGFR) < 30)
3. Patients with malignant tumor, other serious systemic diseases and psychosis.
4. Patients who are participating in other clinical trials or treated with any experimental agents that may contradict this trial (i.e, biologics)
5. Co-Infection of HIV, tuberculosis.
6. Known immunocompromised state or medications known to be immunosuppressive (see concomitant prohibited medications).
7. Intubated patients (due to inability to sign an informed consent)
8. Patients with P/F ratio of <150 or a change in status of eligibility manifested by a rapid decline of P/F ratio between eligibility status and actual drug delivery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of safety by determining the number of participants with any Adverse Events (AE) and Serious Adverse Events (SAE) | 28 days follow up
  Incidence rates and severity of any Adverse Events (AE) and Serious Adverse Events (SAE)

SECONDARY OUTCOMES:
Preliminary Efficacy: Recovery from COVID-19 as determined by negative PCR or asymptomatic by the NIH classification for the severity of illness | 28 days follow up
  Recovery from COVID-19 will be determined by the following measures:
  The percentage of subjects reporting to 'Asymptomatic' by the NIH classification and the number of days to reach this classification, and/or The percentage of subjects negative for SARS-CoV-2 RNA (by PCR) and the number of days for viral clearance (negative PCR results)
Mortality | 28 days follow up
  Incidence rate of Mortality from any cause
Preliminary Efficacy: To assess prevention of respiratory deterioration associated with COVID-19 by measuring the PaO2/FiO2 ratio | On days, 3, 5, 7, 14, and 28 during 28 days follow up
  Respiratory function will be assessed by measuring the ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2).
  Patients with PaO2/FiO2 ratio < 300mmHg are considered severe patients.
  • The PaO2/FiO2 ratio and its change from the baseline value will be measured on days, 3, 5, 7, 14, and 28.
Hospitalization | 28 days follow up
  Cumulative days in the Intensive care unit (ICU) or COVID-19 ICU or COVID-19 department and/or in hospital.
Life support | 28 days follow up
  Number of ventilator-free days.
Clinical status by the new NIH Patient Classification for the severity of illness | 28 days follow up
  Change from baseline of the new NIH Patient Classification for the severity of illness.
Clinical status by NEWS2 | 28 days follow up
  Change from baseline of National Early Warning Score (NEWS2).
Support measurements: percentage of subjects reporting each severity rating on a 7-point ordinal scale | 28 days follow up
  Percentage of subjects reporting each severity rating on a 7-point ordinal scale at day 28 as follows:
  1. Death.
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, not requiring supplemental oxygen.
  6. Not hospitalized, limitation on activities.
  7. Not hospitalized, no limitations on activities.
Support measurements: improvement of severity rating on a 7-point ordinal scale | 28 days follow up
  Time to improvement of one category from admission using this 7-point ordinal scale, as follows:
  1. Death.
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, not requiring supplemental oxygen.
  6. Not hospitalized, limitation on activities.
  7. Not hospitalized, no limitations on activities.
Virus Clearance | Within the 28 days follow up, tested on days 14 and 28
  Evaluation of clearance of the virus using PCR (Negative for SARS-CoV-2 RNA) on days 14 and 28 (if not negative before).
Exploratory: Serum cytokines/chemokines and immunomodulating factors | 28 days follow up
  Serum concentrations (pg/ml) of cytokines, chemokines, complement, hematopoietic growth factors, and other immunomodulating factors (including HMGB1) will be measured before and after the infusion of Allocetra-OTS and periodically throughout 28 days follow up.
Exploratory: complete blood counts | 28 days follow up
  Differential blood counts will be performed before and after the infusion of Allocetra-OTS and periodically throughout 28 days follow up.
Exploratory: Histone and cell-free DNA levels | 28 days follow up
  Histone and cell-free DNA plasma levels will be measured before and after the infusion of Allocetra-OTS and periodically throughout 28 days follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mevorach, MD, Principal Investigator — Hadassah Medical Organization; Peter V van Heerden, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baden LR, Rubin EJ. Covid-19 - The Search for Effective Therapy. N Engl J Med. 2020 May 7;382(19):1851-1852. doi: 10.1056/NEJMe2005477. Epub 2020 Mar 18. No abstract available. PMID 32187463
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Derived] van Heerden PV, Abutbul A, Naama A, Maayan S, Makram N, Nachshon A, Abu Jabal K, Hershkovitz O, Binder L, Shabat Y, Reicher B, Mevorach D. Apoptotic cells for treatment of acute respiratory distress syndrome associated with COVID-19. Front Immunol. 2023 Aug 2;14:1242551. doi: 10.3389/fimmu.2023.1242551. eCollection 2023. PMID 37600829